CLINICAL TRIAL: NCT01964300
Title: Phase II Study of Peginterferon Alfa-2b (Sylatron) for Pediatric Patients With Unresectable or Recurrent Craniopharyngioma
Brief Title: Peginterferon Alfa-2b in Younger Patients With Craniopharyngioma That is Recurrent or Cannot Be Removed By Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy (stratum 2); slow accrual (stratum 1)
Sponsor: Pediatric Brain Tumor Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBTC-039; NCI-2013-01639 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PBTC-039 (Other: Pediatric Brain Tumor Consortium); PBTC-039 (Other: CTEP); U01CA081457 (NIH)
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Childhood Craniopharyngioma
MeSH Terms: interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (peginterferon alfa-2b) (Experimental): Patients receive peginterferon alfa-2b subcutaneously (SC) weekly for 6 weeks. Treatment may repeat every 6 weeks for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: peginterferon alfa-2b; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: peginterferon alfa-2b — Given subcutaneously (SC)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well peginterferon alfa-2b works in treating younger patients with craniopharyngioma that is recurrent or cannot be removed by surgery. Peginterferon alfa-2b may interfere with the growth of tumor cells and slow the growth of craniopharyngioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the 1-year disease stabilization rate associated with the use of Sylatron (peginterferon alfa-2b) in patients with progressive unresectable or recurrent craniopharyngiomas following surgery alone who have not received radiation therapy.

II. To estimate the sustained objective response rate (partial response (PR) + complete response (CR)) to Sylatron in patients with craniopharyngiomas which progress or recur following radiation therapy.

SECONDARY OBJECTIVES:

I. To estimate the response rate in patients with progressive unresectable or recurrent craniopharyngioma treated with Sylatron by study stratum.

II. To estimate the progression-free survival distribution for patients with unresectable or recurrent craniopharyngiomas treated with Sylatron by study stratum.

III. To evaluate the toxicity profile of Sylatron in children with unresectable or recurrent craniopharyngiomas.

IV. To compare the protocol specific disease assessment criteria to MacDonald criteria during the first year of treatment in stratum I and at the time of objective response and progressive disease in both strata.

V. To characterize evidence of WNT pathway activation by immunohistochemistry and MAPK pathway activation by pyrosequencing in resected tumor tissue in patients with craniopharyngiomas, and correlate these results with outcome and response data.

OUTLINE:

Patients receive peginterferon alfa-2b subcutaneously (SC) weekly for 6 weeks. Treatment may repeat every 6 weeks for up to 18 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have a histologically verified diagnosis of craniopharyngioma

  * Stratum 1: patients with progressive unresectable or recurrent craniopharyngiomas treated with surgery alone, who have not received radiation therapy; patients with unresectable craniopharyngiomas, (i.e. residual measurable disease following surgical resection) will be enrolled at the time of progression
  * Stratum 2: patients with progressive or recurrent craniopharyngiomas following radiation therapy
* All patients must have measurable residual disease defined as tumor measurable in two perpendicular diameters on magnetic resonance imaging (MRI)

  * Please note: measurements are required for both the solid and cystic components
* Subjects must have recovered from the acute toxicities of all prior therapy before entering this study; for those acute baseline adverse events attributable to prior therapy, recovery is defined as a toxicity grade =< 2, using Common Terminology Criterial for Adverse Events (CTCAE) version (v.) 4.0, unless otherwise specified in the inclusion and exclusion criteria
* Myelosuppressive chemotherapy (includes intra-cystic bleomycin):

  * Subjects must have received their last dose of known myelosuppressive anticancer chemotherapy at least three (3) weeks prior to study registration or at least six (6) weeks if nitrosourea
* Subjects must have received their last dose of investigational or biologic agent >= 7 days prior to study registration

  * In the event that a subject has received an investigational or biologic agent and has experienced >= grade 2 myelosuppression, then at least three (3) weeks must have elapsed prior to registration
  * If the investigational or biologic agent has a prolonged half-life (>= 7 days) then at least three (3) weeks must have elapsed prior to registration
* Subjects must have completed at least 3 half-life periods from the last dose of monoclonal antibody prior to registration

  * Note: a list of half-lives of commonly used monoclonal antibodies is available on the Pediatric Brain Tumor Consortium (PBTC) website under Generic Forms and Templates
* Stratum 1: patients must not have received radiation therapy
* Stratum 2: patients must have received radiation therapy, including gamma knife or phosphorus-32 (P32)

  * More than 6 months from the time of enrollment if the recurrence is predominantly solid
  * More than 12 months from the time of enrollment if the recurrence is predominantly cystic
* At least 7 days since the completion of therapy with a hematopoietic growth agent (filgrastim, sargramostim, and erythropoietin) and 14 days for long-acting formulations
* Karnofsky performance scale (KPS for > 16 years [yrs] of age) or Lansky performance score (LPS for =< 16 years of age) >= 60 assessed within two weeks prior to registration
* Age: 18 months - 25 years (Minimum weight 20 Kilogram is required to be eligible for the study, since the minimum injection volume of SYLATRON is 0.05 ml, 20 mcg, subcutaneously (SQ) as suggested by Merck)
* Absolute neutrophil count (ANC) >= 1000/ul (unsupported)
* Platelets >= 100,000/ul (unsupported)
* Hemoglobin (Hg) >= 8g/dL (unsupported)
* Alanine aminotransferase (ALT) =< 2.5 x the upper limit of institutional normal
* Total bilirubin =< x 1.5 upper limit of institutional normal
* Serum creatinine =< 1.5 x the upper limit of normal for age, or calculated creatinine clearance or nuclear glomerular filtration rate (GFR) >= 70 ml/min/1.73 m^2

  * =< 0.6 mg/dL (1 to < 2 years of age)
  * =< 0.8 mg/dL (2 to < 6 years of age)
  * =< 1.0 mg/dL (6 to < 10 years of age)
  * =< 1.2 mg/dL (10 to < 13 years of age)
  * =< 1.4 mg/dL (females >= 13 years of age)
  * =< 1.5 mg/dL (males 13 to < 16 years of age)
  * =< 1.7 mg/dL (males >= 16 years of age)
* All patients must have undergone at least one surgical procedure to verify the diagnosis
* Patients must have evidence of radiographic progression as defined below:

  * Stratum 1: defined as >= 25% increase in the product of the greatest perpendicular diameters of the tumor as a whole (solid and cystic component) AND >= 0.4 cm increase in each of at least two dimensions of the tumor as a whole OR any new or worsening neurologic/vision deficit in conjunction with a lesser change in the solid or cystic component
  * Stratum 2:

    * For patients more than 6 months following radiation therapy (RT) (including radiosurgery or P32), progression is defined as a >= 25% increase in the product of the greatest perpendicular diameters of the solid component AND >= 0.4 cm increase in each of at least two dimensions of the solid component
    * For patients more than 12 months following RT (including radiosurgery or P32), progression is defined as >= 25% increase in each of the product of the greatest perpendicular diameters of the solid tumor AND >= 0.4 cm increase in each of at least two dimensions of the solid tumor; patients demonstrating isolated cyst progression more than 12 months after RT must show a continued increase in the cystic component on two serial MRI scans performed at least 4 weeks apart OR re-accumulation of the cyst following one or more cyst aspirations; patients with progressive neurologic signs and/or symptoms associated with isolated cyst formation or progression are eligible if the neurologic signs and/or symptoms do not improve within 4 weeks of cyst aspiration
* Female subjects of childbearing potential must not be pregnant or breast-feeding; female subjects of childbearing potential must have a negative serum or urine pregnancy test; (pregnancy test must be repeated within 72 hours prior to the start of therapy)
* Subjects of childbearing or child fathering potential must be willing to use a medically acceptable form of birth control, which includes abstinence, while being treated on this study
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Stratum 1 patients: must not have had > 3 surgical debulking procedures/resections
* Patients may not have received prior interferon, either systemic or intra-cystic
* Patients must not have evidence of metastatic tumor
* Patients must not be on steroids other than for physiologic replacement
* Patients must not have a severe psychiatric illness, including major depression or any previous suicide attempts
* Patients must not be on phenytoin, warfarin or methadone due to potential drug interactions
* Patients must not have known hypersensitivity reactions, such as urticaria, angioedema, bronchoconstriction, anaphylaxis, Steven-Johnson syndrome, and toxic epidermal necrolysis to interferon alpha or any other products component
* Subjects with inability to return for follow-up visits or obtain follow-up studies required to assess toxicity to therapy

Ages: 18 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stewart Goldman, Principal Investigator — Ann & Robert H. Lurie Children Hospital of Chicago
Locations (9):
- United States (9):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Stanford University and Lucile Packard Children Hospital, Palo Alto, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Lurie Children's Hospital, Chicago, Illinois
  - National Cancer Institute Pediatric Oncology Branch, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Children Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - St. Jude Children Research Hospital, Memphis, Tennessee
  - Texas Children's Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients 18 months to 25 years with histologically confirmed craniopharyngioma were enrolled at Pediatric Brain Tumor Consortium (PBTC) member institutions. The first patient was enrolled on 4/1/2014 and the last patient was enrolled on 11/20/2017. Accrual was halted early due to lack of efficacy in stratum 2 and slow accrual in stratum 1.
Pre-assignment Details: Stratum 1 patients had progressive unresectable or recurrent craniopharyngiomas treated with surgery alone. Stratum 2 patients had progressive/recurrent craniopharyngiomas following radiation. 19 patients were enrolled (7 stratum 1, 12 stratum 2); one of the stratum 2 patients was ineligible leaving 18 eligible patients (7 stratum 1, 11 stratum 2).
Groups:
- Stratum 1: Stratum 1 patients are those with progressive unresectable or recurrent craniopharyngiomas treated with surgery alone, who had not received radiation therapy. Treatment consisted of Peginterferon alfa-2b (Sylatron) subcutaneously weekly for 6 weeks. Treatment may repeat every 6 weeks for up to 18 courses in the absence of disease progression or unacceptable toxicity.
- Stratum 2: Stratum 2 patients are those with patients with progressive or recurrent craniopharyngiomas following radiation therapy. Treatment consisted of Peginterferon alfa-2b (Sylatron) subcutaneously weekly for 6 weeks. Treatment may repeat every 6 weeks for up to 18 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Stratum 1 | Stratum 2
Started | 7 | 12
Completed | 1 | 1
Not Completed | 6 | 11
Not completed — Ineligible after enrollment | 0 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 3 | 5
Not completed — Withdrawal by Subject | 0 | 1
Not completed — To receive alternative therapy | 1 | 2
Not completed — Enlargement of cyst requiring drainage | 1 | 0
Not completed — Weight criteria not met | 0 | 1

BASELINE CHARACTERISTICS:
Population: The one stratum 2 patient found to be ineligible after enrollment was excluded. Summary statistics for baseline characteristics are shown for eligible patients only (n=18).
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 | Stratum 2 | Total
Number analyzed (Participants) | 7 | 11 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 5 | 12
  Between 18 and 65 years | 0 | 6 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 10.6 [2.0 to 17.0] | 20.5 [6.1 to 25.0] | 13.1 [2.0 to 25.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 10
  Male | 3 | 5 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 4 | 8 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 7 | 11 | 18

OUTCOME MEASURES:

1. Primary Outcome: Rate of Disease Stabilization at 1 Year (i.e., 9 Courses of Treatment) (for Stratum 1 Patients Only)
Description: The percentage of stratum 1 patients with disease stabilization at 1 year is reported, along with a 95% exact confidence interval for the estimate of the true 1-year disease stabilization rate.
Time Frame: Up to 1 year
Population: This primary outcome measure only relates to stratum 1 patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 7 | 0
percentage of participants | 28.6 [5.3 to 65.9] |

2. Primary Outcome: Sustained Objective Response (PR+CR) Rate Observed During the First Year of Treatment (for Stratum 2 Patients Only)
Description: Objective responses had to be sustained for 3 months. The percentage of participants with sustained objective responses is reported with an exact 95% confidence interval of the true sustained objective response rate.
Time Frame: Up to 1 year
Population: Only eligible stratum 2 patients are included in this analysis. This is a *secondary* outcome measure for stratum 1 patients and is therefore reported as a separate outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 0 | 11
percentage of participants |  | 0.0 [0.0 to 25.0]

3. Secondary Outcome: Sustained Objective Response (PR+CR) Rate Observed During the First Year of Treatment (for Stratum 1 Patients Only)
Description: as for outcome 2
Time Frame: Up to 1 year
Population: The seven stratum 1 patients are included in this analysis. This outcome measure was a *primary* outcome measure for stratum 2 patients and is therefore reported as a separate outcome measure for stratum 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 7 | 0
percentage of participants | 14.3 [0.01 to 55.4] |

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS estimates for each stratum were estimated using the method of Kaplan and Meier. PFS was defined as the time interval from date on treatment to the earliest date of disease progression, second malignancy, or death; or to date of last contact for patients without events. One- and two-year PFS estimates are reported by stratum. Only eligible patients were included in this analysis (7 stratum 1 patients and 11 stratum 2 patients).
Time Frame: 2 years after treatment start
Population: The one ineligible stratum 2 patient enrolled on the study was excluded from this analysis, leaving 7 stratum 1 patients and 11 stratum 2 patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 7 | 11
percentage of participants
  PFS at 1 year | 83.3 [50.0 to 100.0] | 68.2 [39.8 to 96.6]
  PFS at 2 years | 27.8 [0.0 to 60.5] | 34.1 [0.0 to 72.5]

ADVERSE EVENTS:
Time Frame: Up to 2 years after start of treatment
Description: Adverse events were graded according to the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. All grades 3 through 5 adverse events while on treatment or within 30 days of treatment were to be collected, in addition to grades 1 and 2 adverse events if the attribution was at least possibly related. All adverse events collected and reported in the study database are reported here.
Groups:
- Stratum 2: Stratum 2 patients are those with patients with progressive or recurrent craniopharyngiomas following radiation therapy. Treatment consisted of Peginterferon alfa-2b (Sylatron) subcutaneously weekly for 6 weeks. Treatment may repeat every 6 weeks for up to 18 courses in the absence of disease progression or unacceptable toxicity.
  Since the ineligible patient received 2 days of Peginterferon alfa-2b, that patient is included in all adverse event reporting results.
Arm/Group | Stratum 1 | Stratum 2
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/12
Serious Adverse Events (participants affected / at risk) | 1/7 | 5/12
Other Adverse Events (participants affected / at risk) | 7/7 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 (N=7) | Stratum 2 (N=12)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stratum 1 (N=7) | Stratum 2 (N=12)
Anemia (Blood and lymphatic system disorders) | 3 (3) | 3 (4)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Floaters (Eye disorders) | 0 (0) | 1 (1)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 4 (5)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (2)
Chills (General disorders) | 3 (8) | 0 (0)
Fatigue (General disorders) | 5 (9) | 3 (4)
Fever (General disorders) | 7 (11) | 2 (4)
Flu like symptoms (General disorders) | 0 (0) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (8) | 8 (14)
Alkaline phosphatase increased (Investigations) | 0 (0) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 3 (5) | 10 (15)
Investigations - Other, specify (Investigations) | 2 (2) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (3) | 4 (6)
Neutrophil count decreased (Investigations) | 3 (10) | 8 (18)
Platelet count decreased (Investigations) | 0 (0) | 4 (6)
Weight loss (Investigations) | 4 (5) | 2 (2)
White blood cell decreased (Investigations) | 6 (14) | 8 (12)
Anorexia (Metabolism and nutrition disorders) | 4 (5) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 2 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 6 (8)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (5) | 1 (2)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Abducens nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (5) | 2 (2)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT01964300/Prot_SAP_000.pdf